CLINICAL TRIAL: NCT01316393
Title: Clinical Evaluation of a Salivary Substitute and a Mucoprotective Product on Xerostomia in Head-and-neck Cancer Patients
Brief Title: Effects of Mucoprotective Product on Xerostomia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Camurus AB (Industry)
Collaborators: Liselott Lindh, Principal Investigator, Prosthetic Dentistry, Malmö University, Malmö, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: HS-10-404; NCT01288118 (obsolete NCT alias)
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Xerostomia
Keywords: xerostomia, saliva, mucoprotection, oral health
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- XER2020 (Experimental): mucoprotective product
  Interventions: Other: XER2020
- Saliva Natura (Active Comparator): salivary substitute
  Interventions: Other: XER2020
- XER2020 placebo (Placebo Comparator)
  Interventions: Other: XER2020

INTERVENTIONS:
Other: XER2020 — mucoprotective product

SUMMARY:
In the present study with a randomized, cross-over, blind, placebo controlled design, the effects of a salivary substitute product and a new mucoprotective product with similar mechanisms of action but with different composition and characteristics will be evaluated in cancer patients suffering from xerostomia.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years of age.
2. The patient must have clinical symptoms of xerostomia (dry mouth) due to treatment of head and neck cancer
3. The patient must understand and consent in writing to the procedure.

Exclusion Criteria:

1. Do not meet the criterion for "dry mouth" regarding saliva secretion threshold values.
2. Known allergy to ingredients in the products to be used in the trial and/or allergy to soy, peanuts, citrus fruit,Yerba Santa or methyl parabene
3. Patients who are unable or unwilling to cooperate with study procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
OHIP questionaire health impact profile | 7 days
  Effect on oral health quality will be assessed after each treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Prosthetic Dentistry, Malmö University, Malmo, Sweden